CLINICAL TRIAL: NCT03272009
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the FXR-agonist EYP001a in Chronically HBV Infected Subjects
Brief Title: Evaluation of the Safety and Pharmacology of EYP001 in HBV Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Collaborators: CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EYP001-103; 2017-002211-33 (EudraCT Number)
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Treatment A (Experimental): oral EYP001a
  Interventions: Drug: EYP001a
- Treatment B (Experimental): oral EYP001a
  Interventions: Drug: EYP001a
- Treatment C (Experimental): oral EYP001a
  Interventions: Drug: EYP001a
- Treatment D (Experimental): oral EYP001a
  Interventions: Drug: EYP001a
- Treatment E (Placebo Comparator): oral placebo
  Interventions: Drug: Placebo
- Treatment F (Active Comparator): oral Entecavir
  Interventions: Drug: Entecavir
- Treatment G (Experimental): oral EYP001a plus subcutaneous injection of Peg-INFα2a
  Interventions: Drug: EYP001a; Drug: peg-interferon alfa-2a
- Treatment H (Experimental): oral EYP001a plus subcutaneous injection of Peg-INFα2a
  Interventions: Drug: EYP001a; Drug: peg-interferon alfa-2a
- Treatment I (Placebo Comparator): oral placebo plus subcutaneous injection of Peg-INFα2a
  Interventions: Drug: Placebo; Drug: peg-interferon alfa-2a

INTERVENTIONS:
Drug: EYP001a — Capsules administered orally. Number of morning and evening capsules depending on treatment arm
  Arms: Treatment A; Treatment B; Treatment C; Treatment D; Treatment G; Treatment H
Drug: Placebo — Placebo capsules for oral administration, identical in appearance to the EYP001a capsules
  Arms: Treatment E; Treatment I
Drug: Entecavir — Tablets administered orally
  Arms: Treatment F
Drug: peg-interferon alfa-2a — Ready-to-Use pre-filled syringes for subcutaneous injection
  Arms: Treatment G; Treatment H; Treatment I

SUMMARY:
Bile acids regulating farnesoid X receptor (FXR) interact with hepatitis B virus replication. EYP001a is a selective, synthetic FXR agonist under development for the treatment of hepatitis B.

This Phase 1b study is designed primarily to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of EYP001a in chronically HBV infected subjects.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled two-part trial.

In Part A, EYP001a will be administered as 29 days monotherapy. Three dose-levels and 2 dosing regimens of EYP001a will be explored against placebo. The design also includes an open-label standard of care Entecavir monotherapy arm (comparator). Subjects will be randomly assigned to one of the 6 treatment arms:

* Treatment A: oral EYP001a
* Treatment B: oral EYP001a
* Treatment C: oral EYP001a
* Treatment D: oral EYP001a
* Treatment E: oral placebo
* Treatment F: oral Entecavir

In Part B, EYP001a or placebo will be administered as 29 days combination therapy with the standard of care Peg-IFNα2a. Subjects will be randomly assigned to one of the 3 treatment arms:

* Treatment G: oral EYP001a plus open label Peg-INFα2a administered as subcutaneous injection
* Treatment H: oral EYP001a plus open label Peg-INFα2a administered as subcutaneous injection
* Treatment I: oral placebo plus open label Peg-INFα2a administered as subcutaneous injection

Subjects enrolled in Part A are eligible for participation in Part B.

Participation will include a 40 day screening period, a 29 day treatment period and a 6 day follow-up evaluation period. For subjects who participate in both Parts A and B, a 14 washout period between Parts A and B will be included.

The safety and tolerability of EYP001a will be assessed by evaluating physical examinations, vital signs, ECGs, clinical laboratory parameters, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Have given voluntary written informed consent;
2. Have a documented medical history of chronic HBV infection (within 12 months of screening visit), both results:

   * Documented positive hepatitis B surface antigen (HBsAg) and
   * Documented HBV DNA > 1000 IU/mL
3. Is anti-HBV treatment naive or treatment experienced (see also exclusion criterion #3).
4. Gender: male or female.
5. Age: 18 to 65 years inclusive.
6. Body mass index (BMI): 17.0-35.0 kg/m2 inclusive.
7. Has clinical chemistry, hematology, coagulation and urinalysis tests within normal, allowable limits (with the exception of alanine aminotransferase [ALT]); see inclusion criterion #10); if there is an out of range value, the result must be considered clinically non-significant by the investigator in order to be eligible.
8. Vital signs after at least 5 minutes resting in supine position at screening within the following ranges:

   * systolic blood pressure: between 90 mm Hg and 145 mm Hg
   * diastolic blood pressure: between 45 mm Hg and 90 mm Hg
   * heart rate: between 40 bpm and 100 bpm
9. Have no clinically significant abnormal 12-lead automatic electrocardiogram (ECG) (incomplete right bundle branch block can be accepted) at screening: PR interval between 120 ms -and 210 ms, QRS-duration < 120 ms, QTc-interval (Fridericia's) ≤ 450 msec.
10. ALT at screening ≤ 5 x upper limit of normal (ULN).
11. Agrees to abstain from all medication, including non-prescription and prescription medication for 28 days prior to the Day 1 study visit, except for authorized medications (such as hormonal contraceptives for females, vitamins prescribed per label dosages and paracetamol). On a case-by-case basis, regular co-medication either as defined on the medication exception list or as documented by written approval from the sponsor as acceptable prior to randomization, will not be considered as a deviation from this criterion.
12. At screening, females must be non-pregnant and non-lactating, or of non-childbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1 year post-menopausal [amenorrhea duration of 12 consecutive months); non-pregnancy will be confirmed for all females by a pregnancy test conducted at screening and at follow-up visit.
13. Female subjects of child-bearing potential, with a fertile male sexual partner, should be willing to use adequate contraception from screening until 90 days after the follow-up visit. Adequate contraception is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the subject, is acceptable.
14. Male subjects, if not surgically sterilized, should be willing to use adequate contraception and not donate sperm from the Day 1 visit to the clinical research centre until 90 days after the follow-up visit. Adequate contraception for the male subject (and his female partner) is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the subject is acceptable.
15. At screening, has no recent (<3 months) history of any clinically significant conditions, which, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results.
16. Willingness to abstain from alcohol from 48 hours prior to each study visit to the clinical research centre.

Exclusion Criteria:

1. Employee of a CRO participating in this study or the Sponsor.
2. Has certain or probable compensated liver cirrhosis documented by at least 2 of the following:

   1. Optional assessment: has documented liver histology Metavir score (F4), Ishak >5 or Scheuer (F4)
   2. Mandatory assessment: has presence or history of ascites, spontaneous bacterial peritonitis, esophageal varices, hepatic encephalopathy
   3. Mandatory assessment: platelet count below 90,000/uL within 12 months of screening visit
   4. Optional assessment: positive indirect blood test of APRI or FIB4 or positive direct blood test Fibrosure, Fibrotest, or FibroSpect within 12 months of screening visit
   5. Optional assessment: has positive elastography within 6 months of screening visit (Fibroscan or Shearwave Aixplorer)
   6. Optional assessment: has abnormal liver imaging (CT/US/MRI) consistent with a lobular/nodular liver and cirrhosis or indirect signs of portal hypertension.
3. Subject is HBV treatment experienced AND currently on anti-HBV treatment during the 30 days (or 5 half-lives of the considered anti-HBV drug, whichever is longer) before the first investigational product administration and until the last study visit.
4. Co-infection with active hepatitis C virus (HCV, except for patients with sustained viral response SVR, who can be included).
5. Co-infection with human immunodeficiency virus (HIV) Note: hepatitis D virus (HDV) status is not required for randomization and if not available can be established during the Day 1 visit with baseline PD virology assessments.
6. Receives or plans to receive systemic immunosuppressive or immunomodulating medications (e.g. IFN) during the study or ≤ 4 months prior to the first investigational product administration.
7. Has clinically relevant immunosuppression from, but not limited to immunodeficiency conditions such as common variable hypogammaglobulinemia.
8. Clinical diagnosis of substance abuse during ≤ 12 months prior to screening with narcotics or cocaine or with alcohol (regular consumption > 21 units/week [men] and > 14 units/week [women]; 1 unit = 1⁄2 pint of beer, 25 mL shot of 40% spirit or a 125 mL glass of wine. Expressed in g/day: > 30 g/day [men] and > 20 g/day [women]).
9. Has a positive drug urine screen (cocaine, phencyclidine, amphetamines (incl. methamphetamines), opiates (incl. heroin, codeine and morphine), benzodiazepines, barbiturates, methadone or alcohol screen. Subjects who admit the occasional use of cannabis will not be excluded as long as they are able to abstain from cannabis when they are assessed at study visits.
10. Has any known pre-existing medical or psychiatric condition that could interfere with the subject's ability to provide informed consent or participate in study conduct, or that may confound study findings.
11. Has a history of long QT syndrome.
12. Has a history of clinically significant gastrointestinal disease, especially peptic ulcerations, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Inflammatory Bowel Syndrome, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, or cardiovascular disease or any other condition which, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results.
13. Has participated in any drug study within 40 days prior to the first drug administration in the current study. Note: Part A participation to this study is acceptable and not an exclusion criteria when considering eligibility for Part B, under the condition that follow-up visit of Part A has been completed and no investigational product related SAEs have occurred during Part A.
14. Has an uncontrolled ongoing illness at screening (e.g., active viral infection).
15. Has had major surgery within 30 days prior to the first drug administration, or within 6 months for gastrointestinal surgery prior to the first drug administration.
16. Has a history of relevant drug and/or food allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Type and frequencies of adverse events | Day 1 through Day 35

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of EYP001 | Day 1 through Day 35
Time to reach maximum concentration (Tmax) after EYP001 administration | Day 1 through Day 35
Area under the concentration-time curve from time 0 to last measurable concentration (AUC0-6h) of EYP001 | Day 1 through Day 35
Bile acid precursor C4 (7αhydroxy-4-cholesten-3-one) | Day 1 through Day 35
Fibroblast growth factor 19 (FGF19) | Day 1 through Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Henk W Reesink, MD, Principal Investigator — Academic Medical Centre AMC Amsterdam; Stephan Riordan, Principal Investigator — Scientia Clinical Research Limited Sydney
Locations (9):
- Australia (2):
  - Scientia Clinical Research Limited, Sydney, New South Wales
  - Linear Clinical Research Limited, Perth, Western Australia
- Netherlands (2):
  - Academic Medical Centre (AMC), Amsterdam
  - Erasmus MC, Rotterdam
- Poland (3):
  - Klinika Chorób Zakaźnych I Hepatologii UMB, Bialystok
  - Klinika Chorób Zakaźnych, Kielce
  - HepID, Lublin
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Hospital for Tropical Diseases, Bangkok